CLINICAL TRIAL: NCT03372499
Title: Effect of Diet Management on Incidence of Hepatic Encephalopathy of Patients With Cirrhosis and Variceal Bleeding After Transjugular Intrahepatic Portosystemic Shunt Treatment
Brief Title: Diet Management on Hepatic Encephalopathy of Patients With Variceal Bleeding After Intrahepatic Portosystemic Shunt Creation
Acronym: DM-PTHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Yang (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Li Yang, Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM-PTHE
Record Dates: First submitted 2017-11-08; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy; Diet Management; Transjugular Intrahepatic Portosystemic Shunt
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutritional management group (Experimental): diet management strategy for encephalopathy
  Interventions: Dietary Supplement: diet management strategy for encephalopathy
- control group (No Intervention): Current ordinary guidance for patients after TIPS placement performed by trained nurse in the inpatient department

INTERVENTIONS:
Dietary Supplement: diet management strategy for encephalopathy — diet management strategy for encephalopathy means diet management strategy from the nutritional management consensus of hepatic encephalopathy.
  Arms: nutritional management group

SUMMARY:
Hepatic encephalopathy is a severe complication of transjugular intrahepatic portosystemic shunt (TIPS) treatment in patients with cirrhosis and variceal bleeding. This study is specially designed to explore whether diet management strategy could decrease incidence of encephalopathy after TIPS treatment.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a severe complication of TIPS treatment in patients with cirrhosis and variceal bleeding. The overall incidence of post-TIPS encephalopathy ranges between 10% and 50%, and even the percentage of the new or worsened HE was evaluated up to 13-36%. No approach or medication was evidenced for prophylaxis of post-TIPS encephalopathy, including lactulose and rifaximin. Diet management has been used as an important part of the prophylaxis and treatment strategy for patients with metabolic diseases like diabetes and nephritis, which has drawn increasing interest of clinicians. Nevertheless, there is still no standard consensus or even recommendation for patients after TIPS procedure for now, which worsened malnutrition and affected survival. Thus, this study is specially designed to explore whether diet management strategy, drawn up from the nutritional management consensus of hepatic encephalopathy (ISHEN consensus), could decrease incidence of encephalopathy after TIPS treatment of the patient with cirrhosis and variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* patients with decompensated liver cirrhosis regardless of the etiology
* acute variceal bleeding or with history of variceal bleeding evidenced by endoscopy
* an age between 18 and 75 years old

Exclusion Criteria:

* a total bilirubin level more than 3mg/dL (51.3mmol/L)
* a creatinine level greater than 3 mg/dL(265umol/L)
* severe dysfunction of heart and respiratory system
* pregnancy
* uncontrolled neoplasm
* active systemic infection
* history of any kind of encephalopathy, mental disease, alcohol dependence, or any other status that influence brain function
* diabetes or any other metabolic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hepatic Encephalopathy | 1 year
  incidence of symptomatic hepatic encephalopathy in all stages within 1 year after enrollment

SECONDARY OUTCOMES:
Liver Transplantation-free Survival Rate | 1 year
  survival rate free of liver transplantation within 1 year after enrollment
Incidence of Stent Dysfunction | 1 year
  Narrowing or even complete occlusion of the stent, evidenced by imaging examination and/or upper gastrointestinal endoscopy, with or without clinic symptoms.
Incidence of Portal Hypertension Related Severe Complications | 1 year
  Incidence of severe complications of portal hypertension, especially for failure of control of acute variceal bleeding and clinical significant rebleeding.
Change of Nutritional Status | 1 year
  Human body components analysis, evaluated by score of the Inbody Test.
Change of Quality of Life | 1 year
  Health related quality of life, assessed by score of the widely used questionaire Short Form 36.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Director — Department of Gastroenterology and Hepatology, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators need to discuss with other participants whether or not to share data of the study.

REFERENCES:
- [Background] Rossle M. TIPS: 25 years later. J Hepatol. 2013 Nov;59(5):1081-93. doi: 10.1016/j.jhep.2013.06.014. Epub 2013 Jun 25. PMID 23811307
- [Background] Somberg KA, Riegler JL, LaBerge JM, Doherty-Simor MM, Bachetti P, Roberts JP, Lake JR. Hepatic encephalopathy after transjugular intrahepatic portosystemic shunts: incidence and risk factors. Am J Gastroenterol. 1995 Apr;90(4):549-55. PMID 7717309
- [Background] Routhu M, Safka V, Routhu SK, Fejfar T, Jirkovsky V, Krajina A, Cermakova E, Hosak L, Hulek P. Observational cohort study of hepatic encephalopathy after transjugular intrahepatic portosystemic shunt (TIPS). Ann Hepatol. 2017 Jan-Feb;16(1):140-148. doi: 10.5604/16652681.1226932. PMID 28051803
- [Background] Luo L, Fu S, Zhang Y, Wang J. Early diet intervention to reduce the incidence of hepatic encephalopathy in cirrhosis patients: post-Transjugular Intrahepatic Portosystemic Shunt (TIPS) findings. Asia Pac J Clin Nutr. 2016;25(3):497-503. doi: 10.6133/apjcn.092015.14. PMID 27440683
- [Background] Nardelli S, Gioia S, Pasquale C, Pentassuglio I, Farcomeni A, Merli M, Salvatori FM, Nikolli L, Torrisi S, Greco F, Nicoletti V, Riggio O. Cognitive Impairment Predicts The Occurrence Of Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt. Am J Gastroenterol. 2016 Apr;111(4):523-8. doi: 10.1038/ajg.2016.29. Epub 2016 Mar 1. PMID 26925879
- [Background] Riggio O, Angeloni S, Salvatori FM, De Santis A, Cerini F, Farcomeni A, Attili AF, Merli M. Incidence, natural history, and risk factors of hepatic encephalopathy after transjugular intrahepatic portosystemic shunt with polytetrafluoroethylene-covered stent grafts. Am J Gastroenterol. 2008 Nov;103(11):2738-46. doi: 10.1111/j.1572-0241.2008.02102.x. Epub 2008 Sep 4. PMID 18775022
- [Background] Riggio O, Masini A, Efrati C, Nicolao F, Angeloni S, Salvatori FM, Bezzi M, Attili AF, Merli M. Pharmacological prophylaxis of hepatic encephalopathy after transjugular intrahepatic portosystemic shunt: a randomized controlled study. J Hepatol. 2005 May;42(5):674-9. doi: 10.1016/j.jhep.2004.12.028. PMID 15826716
- [Background] Riggio O, Ridola L, Angeloni S, Cerini F, Pasquale C, Attili AF, Fanelli F, Merli M, Salvatori FM. Clinical efficacy of transjugular intrahepatic portosystemic shunt created with covered stents with different diameters: results of a randomized controlled trial. J Hepatol. 2010 Aug;53(2):267-72. doi: 10.1016/j.jhep.2010.02.033. Epub 2010 Apr 27. PMID 20537753
- [Background] Riggio O, Nardelli S, Moscucci F, Pasquale C, Ridola L, Merli M. Hepatic encephalopathy after transjugular intrahepatic portosystemic shunt. Clin Liver Dis. 2012 Feb;16(1):133-46. doi: 10.1016/j.cld.2011.12.008. Epub 2012 Jan 4. PMID 22321469
- [Background] Yang Z, Han G, Wu Q, Ye X, Jin Z, Yin Z, Qi X, Bai M, Wu K, Fan D. Patency and clinical outcomes of transjugular intrahepatic portosystemic shunt with polytetrafluoroethylene-covered stents versus bare stents: a meta-analysis. J Gastroenterol Hepatol. 2010 Nov;25(11):1718-25. doi: 10.1111/j.1440-1746.2010.06400.x. PMID 21039832
- [Background] Masson S, Mardini HA, Rose JD, Record CO. Hepatic encephalopathy after transjugular intrahepatic portosystemic shunt insertion: a decade of experience. QJM. 2008 Jun;101(6):493-501. doi: 10.1093/qjmed/hcn037. Epub 2008 Apr 25. PMID 18440957
- [Background] Suraweera D, Sundaram V, Saab S. Evaluation and Management of Hepatic Encephalopathy: Current Status and Future Directions. Gut Liver. 2016 Jul 15;10(4):509-19. doi: 10.5009/gnl15419. PMID 27377741
- [Background] Berlioux P, Robic MA, Poirson H, Metivier S, Otal P, Barret C, Lopez F, Peron JM, Vinel JP, Bureau C. Pre-transjugular intrahepatic portosystemic shunts (TIPS) prediction of post-TIPS overt hepatic encephalopathy: the critical flicker frequency is more accurate than psychometric tests. Hepatology. 2014 Feb;59(2):622-9. doi: 10.1002/hep.26684. PMID 24620380
- [Background] Kramer L, Bauer E, Gendo A, Funk G, Madl C, Pidlich J, Gangl A. Neurophysiological evidence of cognitive impairment in patients without hepatic encephalopathy after transjugular intrahepatic portosystemic shunts. Am J Gastroenterol. 2002 Jan;97(1):162-6. doi: 10.1111/j.1572-0241.2002.05441.x. PMID 11808942
- [Background] Abdelsayed GG. Diets in Encephalopathy. Clin Liver Dis. 2015 Aug;19(3):497-505. doi: 10.1016/j.cld.2015.05.001. PMID 26195204
- [Background] Takuma Y, Nouso K, Makino Y, Hayashi M, Takahashi H. Clinical trial: oral zinc in hepatic encephalopathy. Aliment Pharmacol Ther. 2010 Nov;32(9):1080-90. doi: 10.1111/j.1365-2036.2010.04448.x. Epub 2010 Sep 3. PMID 20822500